CLINICAL TRIAL: NCT02664480
Title: Assesment of Salivary Alpha-amylase Levels Before and After Ovulation: A Randomized Controlled Trial
Brief Title: Assesment of Salivary Alpha-amylase Levels Before and After Ovulation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Mustafa Ozturk, Etimesgut Military Hospital Obstetrics and Gynecology, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: Gulhane School of Medicine
Record Dates: First submitted 2016-01-11; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Salivary Amylase
Keywords: Salivary Alpha-amylase; ovulation
MeSH Terms: interventions — Salivary alpha-Amylases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — salivary amylase
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: Reproductive age women with polycystic ovary syndrome and irregular menses (Salivary Alpha-amylase Levels of 3rd and 24th day of menstrual cyclus)
  Interventions: Other: Salivary alpha-Amylases
- control group: Reproductive age women with regular menses (Salivary Alpha-amylase level of 3rd and 24th day of menstrual cyclus)
  Interventions: Other: Salivary alpha-Amylases

INTERVENTIONS:
Other: Salivary alpha-Amylases — Investigators will collect Salivary alpha-Amylases before and after ovulation

SUMMARY:
Investigators aimed to investigate whether there is an association between ovulation and salivatory alpha amylase (sAA) activity in menstrual cycles during a month period in a group of reproductive women.

DETAILED DESCRIPTION:
Saliva is a readily available specimen, which can be collected by noninvasive procedures and contains many hormones, drugs and antibodies of interest in screening and diagnosis. With a salivary specimen, one can collect multiple specimens at the optimum times for diagnostic information. Saliva can be collected in remote sites by unskilled personnel and, is stable at ambient temperatures for several weeks. Because of diurnal and monthly variations, several steroid hormones need multiple samples collected early in the morning or late at night or at the same time every day for a month to give meaningful results. Such collections are often very expensive, inconvenient or impossible to do with blood.

Investigators aimed to investigate whether there is an association between ovulation and salivatory alpha amylase (sAA) activity in menstrual cycles during a month period in a group of reproductive women.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS (study group)
* Reproductive age regular menses women

Exclusion Criteria:

* pregnancy,
* breastfeeding,
* known liver disease,
* alcohol abuse,
* diabetes mellitus,
* smoking
* treatment with oral glucocorticoids
* treatment with hormonal contraceptives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pcos women will included the study population. Because ovulation don't happen.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Changes of Salivary Alpha-amylase activity | 3rd and 24th day of menstrual cyclus
  Saliva samples will be taken 2 times during the menstrual cyclus (3th day and 24th day).

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Öztürk, M.D, Principal Investigator — Etimesgut Military Hospital

IPD SHARING:
Plan to Share IPD: No